CLINICAL TRIAL: NCT01184703
Title: Effects of a Low Glycemic Index Diet on HbA1c and Lipids in Patients With Type I Diabetes
Brief Title: Low Glycemic Index Diet in Patients With Type 1 Diabetes
Acronym: LGID1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Margareta Bensow Bacos, Steno Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GI-project_1
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Glycemic Index Diet; HbA1c; Lipids
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Low GI food — Comparison of carbohydrates in diabetic patients

SUMMARY:
The purpose of this study is to investigate if a low glycemic index diet in comparison with a medium/high glycemic index diet improves the metabolic control in patients with type 1 diabetes.

DETAILED DESCRIPTION:
The glycemic index (GI) was introduced by Jenkins and co-workers in the early 1980s, and is a concept for ranking of carbohydrate foods based on their effect on postprandial glycaemia. A meta-analysis of randomised controlled trials of the effect of low GI diets in the management of diabetes showed a beneficial effect (i.e., a reduction in HbA1c) of low GI versus high GI foods. However, several critical points concerning the GI concept remain, for instance, how to apply it in practical every day life, how to calculate GI in mixed meals, how to find relevant low GI foods, how to ensure compliance to a low GI diet. The most important issue, however, is the fact that studies on the long-term effects of a low GI diet in type 1 diabetes are lacking. In this study, the critical issue of finding palatable low GI foods will be solved in close collaboration with the food industry. This may lead to the development of new commercial products with low GI, which is necessary if low GI diets are to be advocated for diabetics in the future.

Comparison(s): A low glycemic index diet, compared to a medium/normal glycemic index diet.

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetes, durability >5 years
* Age 20-65 years
* Normal weight (BMI 19-26 kg/m2)
* Diabetic treatment with mealtime and bedtime insulin.
* HbA1c ≤10 %
* Informed consent to participate in the study.

Exclusion Criteria:

* Diabetic complications; neuropathy, foot ulcers and/or gastroparesis.
* A known food intolerance of gluten, leguminous plants, nuts or almonds.
* Pregnancy or breast-feeding.
* Concurrent participation in another research study with metabolic effects.
* Previously regular follow-up with a dietician at SDC during the last year.
* Adjustment during the study of medical treatment other than insulin and/or nutritional supplement with metabolic effects.
* Non acceptance of the study diet or food products that are recommended in the study.
* Disability to read and understand the Danish language.
* Unable to receive and/or store the test products.
* Place of residence >1 hr drive from SDC.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months

SECONDARY OUTCOMES:
LDL-cholesterol | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Bensow Bacos, Ch Diet, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark